CLINICAL TRIAL: NCT06074614
Title: Neural Control of Breathing in Parkinson's Disease: an Exploratory Study
Brief Title: Neural Control of Breathing in Parkinson's Disease
Acronym: NEURON-PD
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL84745.091.23
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Respiratory dysfunction; Neural control of breathing; Transcranial magnetic stimulation; Hypercapnic ventilatory response; Respiratory related evoked potential
MeSH Terms: conditions — Parkinson Disease; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkison's disease: Participants with clinically confirmed Parkinson's disease, Hoehn and Yahr stage 1 to 3.
  Interventions: Diagnostic Test: Hypercapnic ventilatory response; Diagnostic Test: Respiratory related evoked potential; Diagnostic Test: Transcranial magnetic stimulation
- Healthy controls: Participants without Parkinson's disease.
  Interventions: Diagnostic Test: Hypercapnic ventilatory response; Diagnostic Test: Respiratory related evoked potential; Diagnostic Test: Transcranial magnetic stimulation

INTERVENTIONS:
Diagnostic Test: Hypercapnic ventilatory response — Control of breathing is predominantly regulated by feedback of the central chemoreceptors. All chemoreceptors are sensitive to changes in partial pressure of carbon dioxide and via acid-base reactions to hydrogen concentration. The hypercapnic ventilatory response test shows the relationship between end-tidal PCO2 and the resulting minute ventilation.
Diagnostic Test: Respiratory related evoked potential — The RREP is a measure of cerebral cortical activity elicited by short inspiratory occlusion or breathing against inspiratory resistive loads and quantifies the initial arrival and further processing of sensory afferent respiratory information in the cortex.
Diagnostic Test: Transcranial magnetic stimulation — Transcranial magnetic stimulation of the diaphragm is an established tool for investigating the cortical excitability related to breathing. TMS will be delivered over the vertex using a magnetic stimulator and a 110mm double cone coil.

SUMMARY:
Breathing is a complex process, which can be controlled through voluntary command or neural control. Parkinson's disease (PD) is a progressive neurological disorder. Many individuals with PD experience respiratory problems, such as coughing difficulties or shortness of breath. Changes in neural control of breathing could be part of the reason of these respiratory problems. This study will measure whether neural control of breathing is impaired in individuals with PD compared to healthy individuals.

DETAILED DESCRIPTION:
Rationale: Parkinson's disease (PD) is a progressive neurological disorder, characterised by loss of dopaminergic neurons. Respiratory dysfunction is common in patients with PD and can lead to pneumonia, which is a common cause of death in PD. However, the exact mechanism of respiratory dysfunction in PD is unknown. The complex process of neural control of breathing may be involved, but this is understudied. This is partly caused by methodological limitations to quantify neural control of breathing. In this study, we will use respiratory neurophysiological methods to determine whether neural control of breathing is impaired in Parkinson's disease. These techniques are hypercapnic ventilatory response, respiratory related evoked potentials and transcranial magnetic stimulation. This study will test the hypothesis that the neural control of breathing is impaired in individuals with PD compared to healthy subjects.

Objective: Primary Objective: To identify disease (Parkinson's disease) specific alterations in neural control of breathing by using respiratory neurophysiological techniques.

Study design: Exploratory cross-sectional study.

Study population: Healthy subjects (n=15) and patients with Parkinson's disease (n=15) >18 years old.

Main study parameters/endpoints:

* Hypercapnic ventilatory response curve (HCVR): HCVR will be determined using the CO2-rebreathing technique.
* Respiratory related evoked potential (RREP): RREP is a measure of cerebral cortical activity elicited by a short inspiratory occlusion.
* Transcranial magnetic stimulation (TMS) diaphragm: TMS is an established tool for investigating the cortical excitability related to breathing.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risk of this study for the participants is negligible. Subjects do not directly benefit from participating in this study. The scientific benefit of this study is to achieve a better understanding of the neural control of breathing in Parkinson's disease. The outcomes of this study may give rise to future new treatments in Parkinson's disease. The burden of the separate study procedures is relatively small: there are no invasive procedures and patients continue their medication as usual. However, the total time of the visit and the collective burden of the experiments may be perceived as strenuous. Therefore, subjects will be explicitly informed about this aspect of the study, and enough breaks will be scheduled in the program.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects: competent adult (>18 years) volunteers
* Patients: adult (<18 years) patients with Parkinson's disease, clinically confirmed by a movement disorder specialised neurologist with Hoehn and Yahr staging 1 to 3
* Willingness and ability to understand nature and content of the study
* Ability to participate and comply with study requirements

Exclusion Criteria:

* Healthy subjects: previous or ongoing diseases of the central nervous system
* Patients: previous or ongoing diseases of the central nervous system, other than Parkinson's disease
* History of or current psychiatric treatment
* History of or current brain surgery or epilepsy, unclusing deep brain stimulation
* Neuromuscular disorders
* Pre-existing pulmonary disease, such as chronic obstructive pulmonary disease, asthma or pulmonary fibrosis
* TMS incompatibility (metal parts in head or neck, skin allergies)
* Implanted cardiac pacemaker or defibrillator, neurostimulator, cochlear implant or medical infusion device
* Large or ferromagnetic metal parts in the head (exept for a dental wire)
* Pregnancy
* Smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants: volunteers. Age- and sex-matched to the participants with Parkinson's disease.
  Participants with Parkinson's disease: recruited through the outpatient registry at the Radboud University Medical Center that have approved contact for research purposes.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Hypercapnic ventilatory response curve | baseline - during the test
  Sensitivity slope of the ventilation increase per unit increase in PetCO2, as measured with a rebreathing technique.
Respiratory related evoked potential | baseline - during the test
  A measure of cerebral cortical activity elicited by a short inspiratory occlusion, expressed in the presence, latency and amplitude of components Nf, P1, N1, P2 and P3.
Transcranial magnetic stimulation | baseline - during the test
  Interstimulus interval curves, using a conditioning stimulus at 80% and a test stimulus at 125%.

SECONDARY OUTCOMES:
FVC | baseline - during the test
  Forced vital capacity.
FEV1 | baseline - during the test
  Forced expiratory volume in 1 second.
MIP | baseline - during the test
  Maximal inspiratory pressure.
MEP | baseline - during the test
  Maximal expiratory pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Jonne Doorduin, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands